CLINICAL TRIAL: NCT04224194
Title: Assessment of Real-life Patient Handling Experience of AVT02 Administered Subcutaneous With an Auto-Injector in Patients With Moderate to Severe Active RA
Brief Title: Auto-injector Real Life Handling in Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVT02-GL-303
Record Dates: First submitted 2019-12-10; First posted 2020-01-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-06

CONDITIONS: RA
Keywords: auto injector pen in RA patients
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional, Single arm to evaluate autoinjector handling (Other): To assess the real-life patient handling experience with the use of an autoinjector in patients with moderate to severe active Rheumatoid Arthritis (RA) who selfinject AVT02 (adalimumab) subcutaneously (SC).
  Interventions: Combination Product: Adalimumab

INTERVENTIONS:
Combination Product: Adalimumab — Combined product as Drug is delivered through an autoinjector pen on which real-life patient handling experience is assessed.

SUMMARY:
To assess the real-life patient handling experience with the use of an autoinjector in patients with moderate to severe active Rheumatoid Arthritis (RA) who self-inject AVT02 subcutaneously (SC).

DETAILED DESCRIPTION:
This is an autoinjector handling study to assess the ability of patients to self-inject AVT02 with the proposed autoinjector in the normal standard of care setting, and to assess the reliability of the proposed autoinjector for AVT02.

On Week 0 (Day 0) eligible patients will be trained by qualified study site personnel (Investigator-led trained injection) following the first injection. The patient will return to the clinic on Week 2 (Day 14) and will be asked to selfinject the second dose (trained self-injection). The injection will be observed by the study personnel and the patient provided any assistance necessary to complete an acceptable injection.

On Week 4 (Day 28), Week 6 (Day 42), and Week 8 (Day 56), the patient will return to clinic and will be asked to self-inject the dose without assistance but under observation of qualified trial staff (observed self-injection).

Observations of autoinjector handling events are recorded independently by both trial site staff and patients using standardized questionnaires.

Any failures to inject will be investigated to determine if they are mechanical failures of the device or due to use error of the patient.

All failures will be further investigated to determine the root cause, and where necessary, appropriate mitigation will be developed and implemented.

In the Extension period (Weeks 9 to 56), AVT02 40 mg will be administered every other week via prefilled syringe (PFS) starting from Week 10 and ending at week 54. The final efficacy evaluation is expected at Week 56.

The clinical study report (CSR) will include the data from the 8week active period. The extension phase CSR will include the data from the 48-week extension period (Weeks 9 to 56).

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, 18 to 80 years of age, inclusive, at time of Screening.
* Patients diagnosed with RA for at least 4 months and currently classified according to the 2010 American College of Rheumatology (ACR)/ European League Against Rheumatism classification criteria for RA (score ≥ 6/10).
* Patients with moderate to severe active RA as defined by ≥ 6 swollen (out of 66) and ≥ 6 tender (out of 68) joint counts and abnormal elevation of C-Reactive Protein (CRP) (≥ 6 mg/L) and fulfills one of the two criteria at screening: a) Positive rheumatoid factor b) Evidence of one joint erosion on radiological assessment of the hands, wrists, or feet at Screening.
* Disease Activity Score in 28 joints C-reactive protein (DAS28 CRP) score of ≥ 3.2 at Screening.
* Eligible to receive treatment on ambulatory care.
* RA functional Class I, II, or III.
* Patients must be taking methotrexate (MTX) orally for ≥ 12 weeks at a stable dose of ≥ 12.5 mg in the last 4 weeks prior to screening and plan to remain on stable dose throughout the study. Patients who are on methotrexate for a minimum of 10 mg per week will be eligible if there is documented intolerance to further dose escalation.
* If patients are using oral corticosteroids, they must have been on a stable dose of up to 10 mg/day prednisolone or equivalent, for ≥ 4 weeks prior to first study dose.
* Naive to adalimumab. Prior treatment with one biologic is allowed.
* Patient has a negative QuantiFERON test for tuberculosis (TB) during Screening.
* Note: Patients with a positive and indeterminate QuantiFERON test are allowed if they have all of the following:
* No evidence of active TB on chest radiograph within 3 months prior to the first dose of study drug.
* Documented history of adequate prophylaxis initiation prior to receiving study drug in accordance with local recommendations.
* No known exposure to active TB after most recent prophylaxis.
* Asymptomatic at Screening and baseline (BL).
* Patients who test positive for TB must be treated for 1 month prior to taking part in the study. Investigators should check with the medical monitor before enrolling patients receiving active treatment for TB.
* Investigators should check with the medical monitor before enrolling such patients.
* Sexually active women of childbearing potential must agree to use highly effective contraception (hormonal contraception pills or injection or implants, sterilization, and abstinence) for the duration of the study and until 3 months after the last dose of the study drug.
* Male patients must agree to use contraception for the duration of the study and agree not to donate sperm during and for 3 months after the last dose of study drug.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legal representative) has been informed of all pertinent aspects of the study.
* Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Patients with previous experience of self-administering medications using an autoinjector or pen (either marketed or investigational).
* Patients who upon initial training are determined not to be acceptable candidates for self-administration.
* RA with significant secondary involvement of any systemic organ (including but not limited to vasculitis, pulmonary fibrosis).
* Prior treatment with more than 1 biologic or 1 protein kinase inhibitor DMARD for RA.
* Previous receipt of HUMIRA® (adalimumab) or a biosimilar of adalimumab.
* Prior treatment with TNF inhibitors for RA with lack of efficacy as per clinical judgment.
* Treatment with DMARD other than MTX within 4 weeks prior to screening (8 weeks in case of leflunomide and azathioprine).
* History of or current inflammatory joint disease other than RA (eg, gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic autoimmune disorder (eg, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease, or any overlap syndrome).
* Any surgical procedure, including bone/joint surgery/synovectomy (including joint fusion or replacement), within 8 weeks prior to informed consent or planned during the study, or history of infected joint prosthesis within 5 years.
* Pregnancy or breast feeding.
* Significant cardiac (eg, New York Heart Association ≥ III) or pulmonary disease (including obstructive pulmonary disease).
* Evidence of clinically significant uncontrolled concomitant disease (cardiac, renal, hepatic, pulmonary, metabolic, or gastro-intestinal) which in the Investigator's or medical monitor's opinion would preclude patient participation.
* Primary or secondary immunodeficiency (history of or currently active), including known history of human immunodeficiency virus (HIV) infection.
* Patient has an active and serious infection or history of infections as follows:
* Any active infection:
* For which non-systemic anti-infectives were used within 4 weeks prior to Day 0 (BL). Note: patients receiving topical antibiotics for facial acne do not need to be excluded.
* Which required hospitalization or systemic anti-infective within 8 weeks prior to Day 0 (BL).
* Recurrent or chronic infections or other active infection that, in the opinion of the Investigator or designee, might cause this study to be detrimental to the patient.
* Invasive fungal infection or mycobacterial infection.
* Opportunistic infections, such as listeriosis, legionellosis, or pneumocystis.
* Patient has a history of malignancy within 5 years except for adequately treated cutaneous squamous or basal cell carcinoma, in situ cervical cancer, or in situ breast ductal carcinoma.
* Any neurological (congenital or acquired), vascular or systemic disorder which could affect any of the efficacy assessments.
* Has evidence (as assessed by the Investigator or designee using good clinical judgment) of active substance abuse (alcohol or drugs) within 6 months of Screening that may impact patient's ability to participate in the study.
* Patient has a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to active substance or to any of the excipients of Humira or AVT02.
* Treatment with any investigational agent 90 days prior to informed consent or 5 halflives of the investigational drug (whichever is longer) and unwilling to undergo washout.
* Previous treatment with any cell-depleting therapies, excluding cyclosporine or MTX, within previous 12 months, including investigational agents. Patients who have received cyclosporine, leflunomide, cyclophosphamide, or azathioprine in the past must have recovered from all drugrelated adverse events (AEs).
* Patient has received live or attenuated vaccines during the 4 weeks prior to Day 0 (BL) or has the intention of receiving a live or attenuated vaccine at any time during the study.
* Intra-articular or parenteral glucocorticoids within 4 weeks prior to informed consent.
* Positive tests for HIV, hepatitis B surface antigen, or hepatitis C serology.
* Hemoglobin < 8.0 g/dL.
* Absolute Neutrophil Count < 1500 cells/mm3.
* Absolute Lymphocyte Count < 800 cells/mm3.
* Platelet count < 100 000 mm3.
* Aspartate aminotransferase and/or alanine aminotransferase that is persistently ≥ 2 × the upper limit of normal. (Persistently indicates at least on 2 occasions separated by a number of days).
* Creatinine clearance < 50 mL/min (Cockcroft-Gault formula).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
percentage of successful self-injections patient rated | up to the Week 8
  The percentage of successful self-injections as reported in the questionnaires completed by the patients (Patient Assessment Tool, Question 1), analyzing all self-injections occurring after the trained self-injection. The higher the % the better the result.
percentage of successful self-injections site staff rated | up to the Week 8
  The percentage of successful self-injections as reported in the questionnaires completed by the trial site personnel (Observer Assessment Tool, Question 1) , analyzing all self-injections occurring after the trained self-injection. The higher the % the better the result.

SECONDARY OUTCOMES:
frequency of any autoinjector handling events during the self-injection process | Up to week 8
  An autoinjector handling event is any event preventing the patient from successfully, selfinjecting the full contents of the autoinjector and occurring after the training selfinjection with the autoinjector pen. The lower the number the better the result.

CONTACTS AND LOCATIONS:
Overall Officials: Nemanja Damjanov, Prof, Principal Investigator — University School of Medicine, Dir. Inst. of Rheumatology, Belgrade
Locations (9):
- Georgia (5):
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - "National Institute of Endocrinology" LTD, Tbilisi
  - JSC "EVEX Hospitals", Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - Georgian Dutch Hospital LLC, Tbilisi
- Ukraine (4):
  - Communal Noncommercial Enterprise "City Clinical Hospital 8" of Kharkiv City Council, Kharkiv
  - SI D. F. Chebotarev Institute of Gerontology NAMS Ukraine, Kyiv
  - Municipal Institution "Zaporozhye City Clinical hospital No.10", Zaporizhzhya
  - CU "Zaporizhzhia Regional Clinical Hospital" ZRC, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.

REFERENCES:
- [Derived] Damjanov N, Kirvalidze N, Kurashvili N, Berti F, Steiger M, Sobierska J, Guenzi E, Otto H, Sattar A, Haliduola HN, Edwald E, Stroissnig H. Assessment of real-life patient handling experience of AVT02 administered subcutaneously via autoinjector in patients with moderate to severe active rheumatoid arthritis: an open-label, single-arm clinical trial, then an extension phase of AVT02 administered with a prefilled syringe. Expert Opin Biol Ther. 2023 Jul-Dec;23(8):781-789. doi: 10.1080/14712598.2022.2131392. Epub 2022 Oct 26. PMID 36205514